CLINICAL TRIAL: NCT03095547
Title: An Open Label Assessment of the Effect of Coadministration of Posaconazole or Pantoprazole on Systemic Exposure of F901318 and the Effect of F901318 on the Single Dose Pharmacokinetics of Tacrolimus and Cyclosporine A in Healthy Male and Female Subjects
Brief Title: Drug/Drug Interactions With F901318
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study no longer required in current format
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Bio-Kinetic Europe, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F901318-01-11-17
Record Dates: First submitted 2017-03-24; First posted 2017-03-29 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — Cyclosporine; posaconazole; Pantoprazole; olorofim; Tacrolimus

STUDY DESIGN:
Intervention Model Description: Three arm parallel group evaluation with fourth arm in series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- F901318 & cyclosporine A & tacrolimus (Experimental): Interaction between cyclosporine A and tacrolimus with F901318
  Interventions: Drug: cyclosporine A; Drug: F901318; Drug: Tacrolimus
- F901318 & posaconazole (Experimental): Interaction between posaconazole and F901318
  Interventions: Drug: Posaconazole; Drug: F901318
- F901318 & pantoprazole (Experimental): Interaction between pantoprazole and F901318
  Interventions: Drug: Pantoprazole; Drug: F901318
- F901318 (Experimental): F901318 alone
  Interventions: Drug: F901318

INTERVENTIONS:
Drug: cyclosporine A — Pharmacokinetic assessment Area Under the plasma concentration: time Curve (AUC) 0-t
  Arms: F901318 & cyclosporine A & tacrolimus
Drug: Posaconazole — Pharmacokinetic assessment AUC 0-tau
  Arms: F901318 & posaconazole
Drug: Pantoprazole — Pharmacokinetic assessment AUC 0-tau
  Arms: F901318 & pantoprazole
Drug: F901318 — Pharmacokinetic assessment AUC 0-tau
Drug: Tacrolimus — Pharmacokinetic assessment AUC 0-t
  Arms: F901318 & cyclosporine A & tacrolimus

SUMMARY:
Study of interactions between F901318 and multiple doses of posaconazole and pantoprazole and single doses of cyclosporine A and tacrolimus in healthy subjects. Pharmacokinetic (PK) profiles, safety and tolerability will be assessed.

DETAILED DESCRIPTION:
Open label randomised parallel group evaluation of three or four dosing schedules over a period of 21 days. Subjects will be randomised into the groups as follows:

1. Cohort A: Pre-treat with tacrolimus 2 mg on day -9 and cyclosporine A 100 mg on Day -3 and obtain pharmacokinetic (PK) curves for both compounds prior to dosing with F901318. Then, F901318 360 mg b.i.d. for 1 or two days followed by 240 mg b.i.d. for 18 or 19 days (Days 2 or 3-20) and 240 mg o.m. on Day 21 (n=12, ideally 6 females minimum 3 females, 6 males, maximum 9 males). Dose again with tacrolimus on Day 9 and with cyclosporine A on day 16 and obtain full PK curves.
2. Cohort B: F901318 360 mg b.i.d. for 1 or 2 days followed by 240 mg b.i.d. for 5 or 6 days. On Day 8, add posaconazole tablets 300 mg b.i.d. followed by 300 mg daily for 6 days (Days 9-14) and decrease F901318 dose to 120 mg daily from Day 8 onwards. On Day 15, discontinue posaconazole but continue F901318 for a further 6 days at a dose of 120 mg daily (Days 15 to 21) (n=12, ideally 6 females, 6 males).
3. Cohort C: F901318 360 mg b.i.d. for one or two days followed by 240 mg b.i.d for 19 days (Day 1-20) and 240 mg o.m. on Day 21. On Day 8, add pantoprazole 40 mg daily for 7 days. On Day 15, discontinue pantoprazole but continue F901318 240 mg b.i.d to day 20 and 240 mg o.m. on Day 21 (n=12, ideally 6 females, 6 males).
4. Cohort D (optional): F901318 for 21 days. Will be conducted, if necessary after completion of cohorts A-C. Dose schedule to be determined on the basis of results from ongoing study F901318-01-06-16 and cohort A of this study but could be up to 480 mg b.i.d for up to three days followed by up to 360 mg bid for 17-19 days and up to 360 o.m. on Day 21 with the objective of achieving and maintaining C12 of 1µg/mL throughout the dosing period (n=12, ideally 6 females, 6 males). The decision to proceed will be taken based on QC'd pharmacokinetic data by the PI and representative(s) of the Sponsor.

Intensive PK evaluations of F901318 and metabolite and concomitant medications will occur as follows:

* Day 1 (F901318 and metabolite alone)
* Day 7 (F901318 and metabolite alone)
* Day 14 (F901318 and metabolite and posaconazole cohort B)
* Day 21 (F901318 and metabolite)

Peak and trough levels of F901318 and metabolite (and posaconazole in cohort B on Days 8-20) will be obtained on intermediate days.

PK curves for tacrolimus will be obtained from Day -9 to Day -3 and from Day 9 to Day 15 (cohort A)

PK curves for cyclosporine A will be obtained from Day -3 to Day 1 (prior to dosing with F901318) and from Day 18 to Day 21 (cohort A)

Adverse events and 12 lead ECGs will be recorded and blood and urine samples will be obtained for safety evaluation throughout.

All subjects will return for a post-study visit 8 to 10 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males and females of any ethnic origin between 18 and 55 years of age and weighing between 60 and 100 kg inclusive.
2. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations
3. Hepatic transaminases must be within normal limits but congenital non haemolytic hyperbilirubinaemia is acceptable.
4. Negative pregnancy test in all females of child bearing potential at screening and Day -1
5. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

1. Female and male subjects who are not, or whose partners have not used for at least three months prior to screening and are not willing to use appropriate contraception during the study and for 3 months after end of dosing.
2. Pregnancy and lactation.
3. For cohort A only, clinically significant infection within the past 6 months or recurring herpes infections within the past 6 months or history of tuberculosis
4. Subjects who have received any prescribed systemic or topical medication within 14 days of the dose administration unless in the opinion of the Investigator and the medical monitor the medication will not interfere with the study procedures or compromise safety
5. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the dose administration (with the exception of vitamin/mineral supplements) unless in the opinion of the Investigator and the medical monitor the medication will not interfere with the study procedures or compromise safety

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under curve 0-t | 21 days
  Area under curve 0-t

SECONDARY OUTCOMES:
Tolerability: Adverse events | 21 days
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: David Bell, MD, Principal Investigator — BioKinetic Europe

IPD SHARING:
Plan to Share IPD: No